CLINICAL TRIAL: NCT07090317
Title: Iparomlimab and Tuvonralimab in Patients With Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma Failed Second-line Treatment:A Prospective, Single Arm, Phase II Trial
Brief Title: Iparomlimab and Tuvonralimab in HNSCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, ren guoxin, Principal Investigator, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-T286
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Iparomlimab and Tuvonralimab (Experimental): The administration regimen of Iparomlimab and Tuvonralimab is: the recommended dose of Iparomlimab and Tuvonralimab is 5mg/kg, intravenous infusion, with a treatment cycle of 21 days. The subjects will continue to receive treatment with Iparomlimab and Tuvonralimab until the termination criteria are met.
  Interventions: Drug: Iparomlimab and Tuvonralimab

INTERVENTIONS:
Drug: Iparomlimab and Tuvonralimab — The administration regimen of Iparomlimab and Tuvonralimab is: the recommended dose of Iparomlimab and Tuvonralimab is 5mg/kg, intravenous infusion, with a treatment cycle of 21 days. The subjects will continue to receive treatment with Iparomlimab and Tuvonralimab until the termination criteria are met.

SUMMARY:
This study is a single center, non-randomized, prospective phase II clinical trial to evaluate the efficacy and safety of Iparomlimab and Tuvonralimab in patients with with recurrent/metastatic head and neck squamous cell carcinoma failed second-line treatment. The participants would receive cetuximab combined with Iparomlimab and Tuvonralimab until termination criteria are met.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years, regardless of gender; Histologically or cytologically confirmed recurrent or metastatic head and neck squamous cell carcinoma (with primary tumor sites in the oropharynx, oral cavity, hypopharynx, and larynx), with clinical or radiological progression after receiving 2 or more lines of anti-tumor systemic therapy in the recurrent or metastatic stage; ECOG performance status of 0 or 1; Expected survival period ≥ 12 weeks; At least one measurable lesion according to RECIST 1.1 criteria. Lesions that have undergone previous radiotherapy can be used as measurable lesions if disease progression occurs; Availability of tumor tissue for PD-L1 detection (paraffin-embedded specimens within 2 years or fresh tumor tissue); For patients with oropharyngeal cancer, the P16 detection status, determined by IHC method;

Normal function of major organs within 2 weeks before treatment, meeting the following criteria:

Bone marrow function: Hemoglobin ≥ 100g/L, white blood cell count ≥ 4.0×10^9/L or neutrophil count ≥ 2.0×10^9/L, and platelet count ≥ 100×10^9/L without blood transfusion or colony-stimulating factor support; Liver function: Serum total bilirubin level ≤ 1.5 times the upper limit of normal, aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 1.5 times the upper limit of normal; Renal function: Serum creatinine level < 1.5 times the upper limit of normal or creatinine clearance rate ≥ 60ml/min, and blood urea nitrogen ≤ 200mg/L; Urinary protein < +; if urinary protein is +, the 24-hour total protein must be < 500mg; Blood glucose: Within the normal range and/or for diabetic patients, blood glucose is controlled in a stable state during treatment; Cardiac function: No myocardial infarction within 1 year; no unstable angina; no symptomatic severe arrhythmia; no cardiac insufficiency; For women of childbearing age, the serum pregnancy test result must be negative within 7 days before the first administration of the trial drug; males with reproductive capacity or females with the possibility of pregnancy must use highly effective contraceptive methods (such as oral contraceptives, intrauterine devices, abstinence, or barrier contraception combined with spermicides) throughout the trial, and continue contraception for 12 months after the end of treatment.

Subjects voluntarily participate in this study, sign the informed consent form, have good compliance, and cooperate with follow-up; Patients whom doctors believe can benefit from the treatment.

Exclusion Criteria:

* Tumors outside the oropharynx, larynx, hypopharynx, or oral cavity; Previous treatment with anti-CTLA-4 drugs; Central nervous system metastasis and/or carcinomatous meningitis; Patients with hearing loss ≥ grade 2 or neuropathy ≥ grade 2 who are currently receiving anti-tumor treatment; Patients who participated in or are participating in other drug/therapy clinical trials within 4 weeks before the first administration of the study drug; Patients who received hematopoietic stimulating factors (such as granulocyte colony-stimulating factor (G-CSF), erythropoietin, etc.) within 1 week before the first administration of the study drug; Positive results of HIV antibody or Treponema pallidum antibody tests;

Patients with active hepatitis B or hepatitis C:

If HBsAg or HBcAb is positive, additional HBV DNA testing is required (with the test result higher than the upper limit of the normal range); If HCV antibody test result is positive, additional HCV RNA testing is required (with the test result higher than the upper limit of the normal range); Active lung diseases (interstitial pneumonia, pneumonia, obstructive pulmonary disease, asthma) or a history of active pulmonary tuberculosis;

Having any uncontrollable clinical problems, including but not limited to:

Persistent or active (severe) infections; Poorly controlled diabetes; Cardiac diseases (New York Heart Association class III/IV congestive heart failure or heart block); The following conditions occurring within 6 months before the first administration: deep vein thrombosis or pulmonary embolism; myocardial infarction; severe or unstable arrhythmia or angina pectoris; percutaneous coronary intervention, acute coronary syndrome, coronary artery bypass grafting; cerebrovascular accident, transient ischemic attack, cerebral embolism; Large amounts of pleural effusion or ascites with clinical symptoms requiring symptomatic treatment; Patients who concurrently used cytochrome P450 3A4 (CYP3A4) inhibitors within one week before screening; A history of stem cell transplantation or organ transplantation; Patients with a history of psychoactive substance abuse who are unable to abstain or a history of mental disorders; Other severe, acute or chronic medical diseases or laboratory test abnormalities that the researcher judges may increase the risks related to study participation or interfere with the interpretation of study results; Patients judged by the researcher to have poor compliance, or other conditions that make them unsuitable for participating in this trial; A history of other malignant tumors within 5 years, except for cured basal cell carcinoma of the skin, cutaneous squamous cell carcinoma, early-stage prostate cancer, and carcinoma in situ of the cervix.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-31 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
objective response rate | 12 months
  ORR was defined as the percentage of participants in the analysis population who have a Complete Response (CR: disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1.

SECONDARY OUTCOMES:
Progression Free Survival | 12 months
  PFS was defined as the time from enrollment to the first documented PD per RECIST 1.1, or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD
overall survival | 12 months
  OS was defined as the time from enrollment to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up.
Number of Participants Experiencing an Adverse Event (AE) | 12 months
  An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition that was temporally associated with the use of the Sponsor's product was also an AE. The number of participants that experienced at least one AE was reported for each treatment arm.

CONTACTS AND LOCATIONS:
Overall Officials: Yue He, M.D., Principal Investigator — the Ninth People's Hospital Affiliated to Shanghai Jiao Tong University School of Medicine
Locations (1):
- the Ninth People's Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China